CLINICAL TRIAL: NCT02411760
Title: Investigation of Diagnostic Improvement Gained Through Optimization of MR Methods for Breast Cancer Detection
Acronym: BCD
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STU 052014-042
Record Dates: First submitted 2015-02-27; First posted 2015-04-08 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Breast Neoplasms
Keywords: MRI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: 3 Tesla Magnetic Resonance Imaging — Assessment of the performance of DWI/ADC measurements alone, and as an adjunct to dynamic contrast enhanced (DCE) MRI in diagnosing/characterizing breast cancer.
  Other Names: Diffusion Weighted Imaging; Dynamic Contrast Enhanced

SUMMARY:
In a single MRI exam on a research scanner, each lesion will be categorized using the BI-RADS MRI score, which utilizes the DCE data alone, and then again using a modified BI-RADS score, which utilizes both DWI and DCE data. The sensitivity and specificity of each approach will be determined using pathology as the gold standard.

DETAILED DESCRIPTION:
MR examinations will be performed on a 3.0 Tesla GE whole-body scanner using an elliptically driven body coil for transmit and a multi-channel bilateral breast coil for receive. The multi-channel coil will consist of 8, 16 or 31 channels. DCE-MRI: DCE-MRI will be carried out using a three-dimensional (3D) turbo fast lowangle gradient echo sequence (TFE) combined with parallel acquisition Sensitivity Encoding (SENSE) technique. The imaging plane will be set in axial plane so that both breasts are included in the images. One image will be acquired before and four images will be acquired after intravenous administration of a standard dose of 0.1 mmol per kg of body weight of Gadavist (Schering AG, Germany) at a rate of 3ml/sec. with subjects in the prone position, breathing normally during the scan. The total scan time for the DCEMRI will be about 8 minutes.

Pharmacokinetic parameters, including the volume transfer constant Ktrans, the fractional volume of extravascular extracellular space of the target tissue ve, and the rate constant kep, will be estimated by fitting a pharmacokinetic model to the time-intensity curves obtained from the DCE-MRI. In this study, the concentration of tracer Ct(t) after bolus injection is assumed to obey the model proposed by Tofts and Kermode (20). DWI-MRI examinations: The DWI acquisition will occur before and/or after contrast enhancement used in DCE imaging. Immediately after the completion of imaging with the 16 (or 31) channel breast coil, the patient will be repositioned replacing the breast coil with an 8 channel breast coil and additional DWI acquisitions will be made. Data for apparent diffusion coefficient assessment on diffusion-weighted imaging will be acquired using a single-shot Echo Planar Imaging sequence in the transverse plane. The DWI protocol will acquire images with up to 16 different b values. Slice dependent shimming will be performed to provide the maximum B0 homogeneity for each slice. The total scan time for the DWI-MRI will be about 5 minutes.

All of the DWI image data from the MRI examinations will be stored on a dedicated HIPPA compliant computer workstation (located in room NE6.114) for analysis. The relevant parameters will be mean ADC and the histogram of ADC in the lesions.

Conductivity imaging: A B1 map and a spin echo image will be acquired for measuring tissue conductivity (21).

The images used for conductivity measurement will be anonymized and sent to the manufacturer for further development of post-processing techniques.

ELIGIBILITY:
Inclusion Criteria:

Women with Breast Imaging-Reporting and Data System (BI-RADS) 4 or 5 Age ≥ 18 years Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

Subjects who have had a needle biopsy of the suspicious area within the last 6 weeks Subjects who have contraindication to contrast enhanced MRI examination.

Contraindications to MRI examinations include:

Medically unstable

* Heart failure
* Unstable angina
* Child bearing
* Lactating Any contraindication per MRI Screening Form (Appendix A attached).
* Implants contraindicated at 3T, pacemakers
* Poorly controlled diabetes
* Body weight greater than 300 pounds
* Claustrophobic Since each patient is receiving a gadolinium based contrast agent intravenously:
* eGFR < 60 mL/min/1.73m2
* Sickle cell disease
* Hemolytic anemia

Subjects must not be pregnant or nursing due to the potential for gadolinium contrast agents to harm fetuses or nursing infants.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the UTSW Breast Imaging Center referred for breast biopsy due to suspicious mammography or ultrasound exams (SOC) with Breast Imaging-Reporting and Data System (BI-RADS) 4 or 5.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic Improvement Gained using an optimized MR Method for Breast Cancer Detection. | Each of 60 patients will have 1 60 minute scan prior to biopsy
  The sensitivity and specificity of breast cancer detection using ADC maps acquired with a 31 channel breast coil and improved B0 shimming will be compared to the sensitivity and specificity of cancer detection using DCE MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lenkinski, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center - Advanced Imaging Research Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided